CLINICAL TRIAL: NCT04257305
Title: A Cross-sectional Study of Venous Thromboembolism Risk Profiles and Prophylaxis in Neurosurgical Inpatients
Brief Title: Study of Venous Thromboembolism Risk Profiles and Prophylaxis in Neurosurgical Inpatients
Acronym: VTE
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Shengqing Li, Chief Physician,Professor, Huashan Hospital
Other Study IDs: KY2016-396
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Venous Thromboembolism
Keywords: Venous thromboembolism; deep venous thrombosis; neurosurgery; pulmonary embolism
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thromboembolism (VTE), comprising deep venous thrombosis (DVT), pulmonary embolism (PE), or both, is a life-threatening complication in postoperative patients. VTE has been estimated an incidence ranged from 79 per 100000 to 269 per 100000 population1. The incidence of VTE rises up to 3.0% in average among all postoperative neurosurgical patients in recent studies, but the number varies in a large range according to primary diseases. This cross-sectional study was aimed to investigate the incidence, associated risk factors, prophylaxis, treatment, and outcomes of VTE in a large clinical neurosurgery center in China.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), comprising deep venous thrombosis (DVT), pulmonary embolism (PE), or both, is a life-threatening complication in postoperative patients. This cross-sectional study was aimed to investigate the incidence, associated risk factors, prophylaxis, treatment, and outcomes of VTE in a large clinical neurosurgery center in China. 9010 patients underwent neurosurgery procedure were included. Distribution of age, sex, whether received PICC during perioperative period, and some special primary diseases are significantly different between VTE and non-VTE patients. Student's test and chi-square test were performed for analyses. We investigated VTE incidence, risk factors, prophylaxes, treatment and outcomes in postoperative neurosurgical patients, and summarized the VTE susceptible population of the patients, providing a VTE patient profile for neurosurgeons to concern.

ELIGIBILITY:
Inclusion Criteria:

Neurosurgical Inpatients. Underwent neurosurgery procedure.

Exclusion Criteria:

Acute or chronic respiratory failure. Acute myocardial infarction or other serious heart diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 9010 patients underwent neurosurgery procedure were included from Jun 1, 2018 to Dec 31, 2019 in Huashan Hospital. Clinical data about demographic information, VTE incidence, primary diseases, laboratory indexes, treatment, and outcomes were collected.
Sampling Method: Non-Probability Sample
Enrollment: 9010 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of VTE occurrence | 19 months
  VTE incidence in postoperative neurosurgical patients during inhospital time from Jun 1,2018 to Dec 31,2019

SECONDARY OUTCOMES:
Rate of complete vessel recanalization | 19 months
  Complete vessel recanalization rate in postoperative neurosurgical patients during inhospital time from Jun 1,2018 to Dec 31,2019
Rate of partial vessel recanalization rate | 19 months
  Partial vessel recanalization rate in postoperative neurosurgical patients during inhospital time from Jun 1,2018 to Dec 31,2019
Rate of bleeding events | 19 months
  Bleeding events occurred in patients during VTE treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shengqing Li, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital,Fudan university, Shanghai, Shanghai Municipality, China